CLINICAL TRIAL: NCT02826824
Title: BECOME CHILDREN OF HOLDERS Corpus Callosum Agenesis Screened IN PERIOD Antenatal
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6268
Record Dates: First submitted 2016-06-16; First posted 2016-07-11 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Corpus Callosum Agenesis
Keywords: corpus callosum agenesis; agenesis; corpus callosum
MeSH Terms: conditions — Agenesis of Corpus Callosum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The corpus callosum agenesis is an interesting malformation between 0.05% and 1.5% of the general population. This malformation is mostly diagnosed prenatally by ultrasound, usually at 22 weeks of gestation, and the use of prenatal advice is routinely offered to the couple.

Several studies in recent years have helped to define the determinants of prognosis for the unborn child suffers from agenesis of the corpus callosum, whether total or partial. These, mainly retrospective, demonstrated that the isolated nature of the deformity (defined as no other brain malformations and brain extra, absence of abnormal karyotype, maternal poisoning or viral seroconversion when pregnancy) is associated with favorable developments in terms of psychomotor development in 80% of cases Similar results were also found in prospective studies, while the associated nature of the defect seems most heavily encumber the prognosis as other malformation or syndrome associated with agenesis of the corpus callosum Although these recent data have already significantly influence prenatal counseling and outcome of pregnancy, questions about the future of the child carrying a prenatal diagnosis of agenesis of the corpus callosum are still valid.

ELIGIBILITY:
Inclusion criteria:

* Children born between January 2000 and January 2013 carrying a corpus callosum agenesis detected prenatally via the multidisciplinary center for prenatal diagnosis (CPDPN) of the Alsace-Lorraine region,
* Children whose holders of parental authority does not oppose the use of clinical data from their child for research purposes

Exclusion criteria:

* Children whose holders of parental authority are opposed to the use of clinical data from their child for research purposes

Max Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The becom of children with agenesis of the corpus callosum detected prenatally in the Alsace-Lorraine region since January 2000
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
questionnaire | since January 2000 to january 2016

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LAUGEL, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Pediatrie 1 - Hopital de Hautepierre, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No